CLINICAL TRIAL: NCT00125840
Title: A Phase I and Pharmacokinetic Study of Clofarabine in Adult Patients With Advanced Solid Tumors
Brief Title: Clofarabine in Adult Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Organization: Sanofi (Industry)
Other Study IDs: CLO151
Record Dates: First submitted 2005-07-29; First posted 2005-08-02 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Solid Tumors; Leukemia, Lymphocytic, Acute, Pediatric; Leukemia, Lymphocytic, Acute, Adult; Leukemia, Myelocytic, Acute, Pediatric; Leukemia, Myelocytic, Acute, Adult; Myelodysplastic Syndromes, Adult
Keywords: CLO151; Clolar; Pediatric ALL and AML; Adult ALL and AML and MDS
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Clofarabine; Dosage Forms

INTERVENTIONS:
Drug: clofarabine (IV formulation)

SUMMARY:
Clofarabine (injection) is approved by the Food and Drug Administration (FDA) for the treatment of pediatric patients 1 to 21 years old with relapsed acute lymphoblastic leukemia (ALL) who have had at least 2 prior treatment regimens.

This research study of clofarabine will be used for advanced cancer in persons in which drugs are no longer effective or no reliable effective treatment is available. The purpose of this study is to find the answers to the following research questions:

1. What is the largest dose of clofarabine that can be safely administered as an IV infusion (over at least 2 hours) once a week for 3 weeks (days 1, 8 and 15) followed by 1 week of rest and repeated every 28 days?
2. What are the side effects of clofarabine when given on this schedule?
3. How much clofarabine is in the blood at specific times after administration and how does the body get rid of the drug? Once the MTD/RP2D is established, patients will be enrolled at the MTD/RP2D regardless of the PK data with cardiac assessments done every other cycle.
4. Will clofarabine help treat a specific cancer?

ELIGIBILITY:
Inclusion Criteria:

* Have a pathologic diagnosis of advanced solid tumors
* After MTD is established, patients must have a measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Be greater than or equal to 18 years old
* Not eligible for therapy of higher curative potential
* Have a Karnofsky Performance Status (KPS) greater than or equal to 70
* Have an estimated life expectancy of greater than or equal to 12 weeks
* Have a negative serum or urine pregnancy test within 7 days of study enrollment (if patient is a female of childbearing potential)
* Male and female patients who are fertile must agree to use an effective barrier method of birth control (latex condom, diaphragm, cervical cap, etc.) to avoid pregnancy
* Sign a written informed consent form
* Able to comply with study procedures and follow-up examinations
* Have adequate organ function as indicated by the following laboratory values, obtained within 2 weeks prior to registration: ANC: greater than or equal to 1.5 × 10 9th/L; Platelets: greater than or equal to 100 × 10 9th/L; Serum bilirubin: less than 2.0 mg/dL; AST and ALT: less than 3 x ULN (Institutional Upper Limit of Normal) without liver involvement OR less than 5 x ULN(*) with liver involvement; Serum creatinine: less than 2.0 mg/dL; Echocardiogram shortening fraction: greater than or equal to 28%(Not on pharmacologic support); or Ejection fraction greater than or equal to 50% (Not on pharmacologic support).

Exclusion Criteria:

* Received previous treatment with clofarabine.
* Have an active, uncontrolled systemic infection considered opportunistic, life threatening, or clinically significant at the time of treatment.
* Prior malignancy with less than a 2-year disease-free interval, except for adequately treated basal cell or squamous cell skin cancer; or in situ cancer of the cervix.
* Are pregnant or lactating.
* Have a psychiatric disorder(s) that would interfere with consent, study participation, or follow-up.
* Have received any chemotherapy, major surgery, or irradiation, whether conventional or investigational, < 4 weeks before enrollment in this study (6 weeks for mitomycin-C or nitrosourea) and/or have not recovered from acute toxicities of all previous therapy prior to enrollment.
* Have any other severe concurrent disease, which, in the judgment of the investigator, would make the patient inappropriate for entry into this study (eg, uncontrolled severe insulin-dependent diabetes, uncontrolled hypertension, transient ischemic attacks, uncontrolled symptomatic coronary artery disease, etc.).
* Have received prior radiation therapy to greater than or equal to 25% of the bone marrow (eg, no whole pelvic irradiation is allowed) and have not recovered from the acute side effects of radiotherapy.
* Have received prior radiation therapy to the mediastinal region.
* Have a broncho-alveolar pattern evident on chest x-ray.
* Have symptomatic or untreated central nervous system (CNS) metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-08; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD)/recommended phase II dose (RP2D) is the dose at which less than or equal to 1 of 6 patients experience a dose limiting toxicity (DLT) with the next higher dose having at least 2 of 3 or 2 of 6 patients experiencing a DLT.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Mary Crowley Medical Research Center, Dallas, Texas
  - US Oncology Tyler Cancer Center, Tyler, Texas